CLINICAL TRIAL: NCT02501915
Title: Kinesio Taping Effects Applied With Different Directions and Tensions on Electromyography, Electroencephalography, Local Temperature and Muscle Strength
Brief Title: Kinesio Taping Effects Applied With Different Directions and Tensions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Estadual de Goiás (Other)
Collaborators: University of Brasilia (Other)
Responsible Party: Principal Investigator, Thiago Vilela Lemos, Physical Therapy Professor at Universidade Estadual de Goias; Phd Student at Universidade de Brasília, Universidade Estadual de Goiás
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26582214.4.0000.5289
Record Dates: First submitted 2014-02-12; First posted 2015-07-17 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: MYOSITIS
Keywords: Muscle
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinesio Taping (GROUP A) (Experimental): Received the application of KT from muscle Origin to Insertion
  Interventions: Device: Kinesio Taping
- Kinesio Taping (GROUP B) (Experimental): received the application of KT from muscle Insertion to Origen
  Interventions: Device: Kinesio Taping

INTERVENTIONS:
Device: Kinesio Taping — Group A received the application of KT from muscle Origin to Insertion and group B Insertion to Origin, with both groups taped the nondominant limb and the dominant limb was used as control group. Diferent tensions will be applied with the tape to see its possible different affect in the outcomes.
  Other Names: Kinesio Tex Tape FP (Finger Print)

SUMMARY:
The Kinesio Taping (KT ) method was developed more than thirty years ago in order to cause sensory effects through the epidermis and dermis, generating a variety of physiological effects in other systems. Clinical effects are well known levels in muscle, neurological system, injuries, inflammation, edema, among other physiological effects are thus largely in the theoretical framework. Objectives: The aim of this study is to evaluate the Electromyographic (EMG), Electroencephalographic (EEG), muscle temperature and flexibility effects with the Rectus Femoral muscle KT application. Methods: This is a pilot study with six subjects in which they were divided into two groups, A and B. Group A received the application of KT from muscle Origin to Insertion and group B Insertion to Origin, with both groups taped the non-dominant limb and the dominant limb was used as control group. The first application was conducted at 0% and the second with 75 to 100% tension. Evaluations were performed before the first application, immediately and 24 hours later. After this last evaluation, was withdrawn taping, evaluated without taping, reapplied 75 to 100 % of rated voltage and in sequence. The sixth last review was conducted 24 hours after this last application. Before every application a specific vibration was performed on the patellar tendon in order to trigger a neurophysiological imbalance rectus femoral.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have authorized the evaluation procedure and through the Term Informed Consent;
* Individuals male and female of any race, duly enrolled in some college course of Universidade Salgado de Oliveira aged between 18-50 years old;
* Healthy subjects without disorders of locomotion without injury history the last 6 months in the lower limbs.

Exclusion Criteria:

* They are considered unfit for research individuals who do not meet the requirements listed above ;
* Individuals who have higher body mass index (BMI ) to 24.99, as the concentrated presence of fat on muscles can limit the effect of bracing;
* Individuals with musculoskeletal disorders and referring pain. Since there report that the pain and dysfunction of movement restricted range of motion and function muscular18 ;
* Individuals who possess too much on the thigh in which prevent proper attachment of bracing and the EMG electrode , or who refuse to perform the trichotomy .
* they show taping allergy ( an allergy test by putting a small bandage on the skin will be held and observed for 24 hours ) ;
* Patients with any contraindication how physical activity according to the guideline of the American College of Sports Medicine (ACSM , 1995), nerve root involvement, cardiorespiratory conditions and pregnancy .

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Muscle Activity | The outcome will be evaluated 24 hours after the intervention
  Group A (n= 15) received the application of KT from muscle (Rectus femoral) Origin to Insertion, Group B (n= 15) from insertion to origin at the non dominant limb, and the dominant limb will be used as control group. The Eletromiography/ EMG (mV) will be measure during an maximum isometric voluntary contraction.

SECONDARY OUTCOMES:
Neurologic Activity | The outcome will be evaluated 24 hours after the intervention
  Group A (n= 15) received the application of KT from muscle (Rectus femoral) Origin to Insertion, Group B (n= 15) from insertion to origin at the non dominant limb, and the dominant limb will be used as control group. The Eletroencephalography - EEG (Hz) will be measure during an maximum isometric voluntary contraction. Will be analyzed 8 channels related with the motor activity located between the frontal and the central lobe.

OTHER OUTCOMES:
Muscle Stregth | The outcome will be evaluated 24 hours after the intervention
  Group A (n= 15) received the application of KT from muscle (Rectus femoral) Origin to Insertion, Group B (n= 15) from insertion to origin at the non dominant limb, and the dominant limb will be used as control group. The strength will be measure by a Hand Hold Dynamometer (Kg/F) during an maximum isometric voluntary contraction.
Local Temperture | The outcome will be evaluated 24 hours after the intervention
  Group A (n= 15) received the application of KT from muscle (Rectus femoral) Origin to Insertion, Group B (n= 15) from insertion to origin at the non dominant limb, and the dominant limb will be used as control group. The temperature will be measure using Thermography (Degrees Celsius) before the KT applications, and 24 hs after staying with the KT applied to the skin.

CONTACTS AND LOCATIONS:
Overall Officials: João V Matheus, PHD, Study Chair — Universidade de Brasilia

REFERENCES:
- [Derived] Lemos TV, Junior JRS, Santos MGRD, Rosa MMN, Silva LGCD, Matheus JPC. Kinesio Taping effects with different directions and tensions on strength and range of movement of the knee: a randomized controlled trial. Braz J Phys Ther. 2018 Jul-Aug;22(4):283-290. doi: 10.1016/j.bjpt.2018.04.001. Epub 2018 Apr 14. PMID 29728298